CLINICAL TRIAL: NCT06870760
Title: Pre-malignant States to Hematologic Malignancies in Firefighters
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00124175; LCI-LEU-FF-CHIP-001 (Other: Atrium Health)
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Clonal Hematopoiesis of Indeterminate Potential; Monoclonal Gammopathy; Non Hodgkin Lymphoma; Leukemia; Multiple Myeloma; Plasma Cell Disorder
Keywords: Firefighters; CHIP; MGUS
MeSH Terms: conditions — Paraproteinemias; Lymphoma, Non-Hodgkin; Leukemia; Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Blood Cell Count; Clonal Hematopoiesis; Chromatin Immunoprecipitation Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Buccal swabs, whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Firefighter: Participants employed by the Charlotte Fire Department (CFD) with at least 5 years of on-the-job experience between the ages of 40 and 49
  Interventions: Other: Monoclonal Gammopathy; Other: Complete Blood Count with differential (CBC w/ diff); Other: Clonal hematopoiesis (CHIP)

INTERVENTIONS:
Other: Monoclonal Gammopathy — Whole blood will be collected at the Baseline visit to evaluate for monoclonal gammopathy through SPEP, immunofixation, and free light chains.
Other: Complete Blood Count with differential (CBC w/ diff) — Whole blood will be collected at the Baseline visit for CBC with differential which may inform a diagnosis of a plasma cell disorder or other hematological disorder.
Other: Clonal hematopoiesis (CHIP) — Whole blood will be collected at the Baseline visit to be evaluated using next generation sequencing (NGS) detection of CHIP. Deep NGS to identify mutations associated with myeloid neoplasms and CHIP will be performed using an error-correcting next generation sequencing multi-gene panel targeting genes most frequently mutated in CHIP.

SUMMARY:
The purpose of the study is to evaluate if firefighter exposure to hazardous compounds will increase the incidence of premalignant hematological states which subsequently increases the risk of the development of hematologic malignancies, and potentially other pathophysiological consequences.

DETAILED DESCRIPTION:
Firefighters from the Charlotte Fire Department, ages 40-49 and with at least 5 years on the job experience will be offered consent for this study. Consented and eligible participants will have labs collected at the Baseline visit to evaluate for CHIP and monoclonal gammopathy. Buccal swabs (also collected at Baseline) and any remaining blood from the Baseline labs will be collected from participants who consent to collection and banking of their samples for future research. Participants will also complete the Firefighter History Assessment at Baseline.

If clonal hematopoiesis (CHIP) results are interpreted by the investigator as abnormal, the participant will be given a clinical referral if indicated for discussion of diagnosis, potential further diagnostic tests, and implications per standard CHIP management guidelines. If monoclonal gammopathy or other (concerning) abnormality of the complete blood count is detected, the participant will be provided a referral for a clinic visit for diagnostic assessments and followed up per standard of care.

If the participant proceeds with the referral and diagnostic work-up, the final diagnosis (if any) resulting from the initial diagnostic assessment(s) will be collected

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information.
2. Age ≥ 40-49 years at the time of consent (self-reported)
3. Ability of the participant to understand and comply with study procedures for the entire length of the study
4. Currently employed by Charlotte Fire Department (CFD) with at least 5 years on-the -job experience (self-reported)

Exclusion Criteria:

Anyone with a current diagnosis of a hematologic malignancy will be excluded.

Ages: 40 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Firefighters ages 40-49 years old, currently employed by Charlotte Fire Department (CFD) with at least 5 years on the job experience (self-reported)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Clonal Hematopoiesis (CHIP) | From enrollment to availability of lab results, approximately 6 months
  The presence of positive somatic mutation will be determined for each enrolled participant as a binary variable indicating if the participant is harboring clonal hematopoiesis.

SECONDARY OUTCOMES:
Monoclonal Gammopathy (MGUS) | From enrollment to availability of lab results, approximately 1 week
  The presence of monoclonal gammopathy will be determined for each enrolled participant as a binary variable defined as abnormal SPEP, IFE, or FLC result.
Targeted Diagnoses Rate | up to 12 months after all labs have resulted
  The presence of a diagnosis(es) based off standard of care diagnostic assessment(s) will be determined for each enrolled participant and for each diagnosis. Targeted diagnoses: MGUS, Smoldering Multiple Myeloma, Multiple Myeloma, AL Amyloidosis, Other Plasma Cell Disorder, Myelodysplastic Syndrome (MDS), Acute Myeloid Leukemia (AML), Aplastic anemia, Clonal cytopenia of undetermined Significance (CCUS), and Other.
Baseline Survey Results | Baseline
  Baseline survey results will be summarized descriptively. The survey is an 18-item survey collecting data including: demographic information, personal and family health history, social behaviors, firefighting experience, prior history of cancer and other items related to firefighting experience. The survey question responses will be collected as either quantitative responses, nominal categorical responses, or ordered categorical responses.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Druhan, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No